CLINICAL TRIAL: NCT05843760
Title: the Prevalance of Headache and Effects on Biopsychosocial Status in Undergraduate Students
Brief Title: Headache in Undergraduate Students and Biopsychosocial Status
Status: Completed | Type: Observational
Sponsor: şeyda öztürk (Other)
Responsible Party: Sponsor-Investigator, şeyda öztürk, Physiotherapist (also a student in Graduate School of Health Sciences), Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: Hacettepe univercity
Record Dates: First submitted 2023-04-14; First posted 2023-05-06 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Headache Disorders, Primary; Prevalence; Migraine; Student; Psychosocial Problem
Keywords: headache; biopsychosocial; migraine; psychosocial
MeSH Terms: conditions — Headache Disorders, Primary; Migraine Disorders; Headache | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- undergraduate students: Hacettepe University Faculty of Physical Therapy and Rehabilitation undergraduate students
  Interventions: Other: personal information form; Other: headache-specific questionnaires; Other: Questionnaires for assessing biopsychosocial status

INTERVENTIONS:
Other: personal information form — undergraduate student(participants) will be asked; age, weight, height, smoking and alcohol use, and headache.
Other: headache-specific questionnaires — ıd migraine test, numeric rate scale, hit-6 headache impact test, headache information form
Other: Questionnaires for assessing biopsychosocial status — hospital anxiety depression, Discomfort Intolerance Test, pittsburgh sleep quality index, fatigue severity scale, self compassion scale, Body Awareness Questionarre, cervical range of motion, İnternational Physical Activity Questionnaire, 12-Item Short-Form Health Survey

SUMMARY:
The primary aim of this study was to determine the prevalence of headache in undergraduate students. The frequency, duration, localizations and symptoms of headache will be determined with the information obtained as a result of the forms filled in by the participants.

The second aim of this study is to examine the effects of headache on physical, social and psychological status in undergraduate student(participants) from a biopsychosocial perspective.

DETAILED DESCRIPTION:
Headache is one of the most common nervous system disorders in society. 95 percent of the population has experienced a headache at least once in their life. The one-year prevalence is almost 1 in 2 people.

The prevalence of headache increases with age. While there is no difference between the sexes in terms of incidence before adolescence, it is more common in the female population in the post-adolescent period.

The ICF model, developed by the World Health Organization, adopts the biopsychosocial approach to provide a holistic perspective. According to this approach, it is aimed to develop interventions by evaluating and examining the biological and psychosocial effects of illness and disability, functionality, needs and demands of the individual.

Headache is also a disease that should be addressed from a biopsychosocial perspective.

Therefore, the primary aim of this study was to determine the prevalence of headache in undergraduate students. The frequency, duration, localizations and symptoms of headache will be determined with the information obtained as a result of the forms filled in by the participants.

The second aim of this study is to examine the effects of headache on physical, social and psychological status in undergraduate student(participants) from a biopsychosocial perspective.

ELIGIBILITY:
Inclusion Criteria:

* Having undergraduate education at Hacettepe University Faculty of Physical Therapy and Rehabilitation.
* be over 18 years old.
* To know Turkish.
* Volunteer to participate in the study.

Exclusion Criteria:

* Being over 65 years old.
* Having any neurological problem except headache.
* Any additional problems that prevent him from completing the questionnaires and scales.

to be

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: undergraduate students
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
prevelance | april 2023-may 2023
  Headache prevalence in undergraduate students

SECONDARY OUTCOMES:
effect of headache on biopsychosocial status | april 2023-may 2023
  Sleep Quality- Pittsburgh Sleep Quality Index- A minimum of 0 and a maximum of 21 points can be obtained from this scale. The higher the score, the worse the sleep quality.
effect of headache on biopsychosocial status | april 2023-may 2023
  Anxiety Depression Level- Hospital Anxiety Depression Scale- A minimum of 0 and a maximum of 42 points can be obtained from this scale. The higher the score, the higher the severity of anxiety depression.
effect of headache on biopsychosocial status | april 2023-may 2023
  Personal Information Form- In this form, participants' height, weight, age, gender, smoking and alcohol use, whether they have a headache or not, and their education level are questioned. there is no minimum or maximum value
effect of headache on biopsychosocial status | april 2023-may 2023
  Self Compassion- Self Compassion Scale- A minimum of 24 and a maximum of 130 points can be obtained from this scale. The higher the score, the higher the level of self-compassion.
effect of headache on biopsychosocial status | april 2023-may 2023
  Fatigue Level- The Fatigue Severity Scale - A minimum of 0 and a maximum of 9 points can be obtained from this scale. The higher the score, the higher the severity of fatigue.
effect of headache on biopsychosocial status | april 2023-may 2023
  Body Awareness- Body Awareness Scale- A minimum of 18 and a maximum of 126 points can be obtained from this scale. The higher the score, the higher the body awareness.
effect of headache on biopsychosocial status | april 2023-may 2023
  Physical Activity Level- International Physical Activity Questionnaire - The scale score is defined in 3 different categories as a result of the scores obtained in the range of minimum 0 and maximum +3000 points. As the score obtained from the scale increases, the level of physical activity increases. results are reported in categories. (low activity levels, moderate activity levels, or high activity levels).
effect of headache on biopsychosocial status | april 2023-may 2023
  Cervical Range of Motion- The participant is asked to evaluate the cervical joint range of motion in 6 directions (flexion, extension, right/left lateral flexion, and right/left rotation). The minimum score is 0, the maximum score is 10. The higher the score, the higher the range of motion.
effect of headache on biopsychosocial status | april 2023-may 2023
  Quality of Life-Short Form-12 (SF-12) - The total score ranges from 0-100. The higher the score, the higher the quality of life.
effect of headache on biopsychosocial status | april 2023-may 2023
  Discomfort intolerance level- Discomfort Intolerance Scale- The total score changes from a minimum of 0 to a maximum of 42 points. As the total scores of the participants increase, it is accepted that the tolerance to the discomfort is higher.
effect of headache on biopsychosocial status | april 2023-may 2023
  Numeric Rate Scale- A minimum of 0 and a maximum of 10 points is obtained from the scale. A high score indicates a high headache.
effect of headache on biopsychosocial status | april 2023-may 2023
  ID- MIGRAINE TEST-There are 3 questions in this test. It is stated that the participants who answer yes to two of the questions are more likely to have migraine.
effect of headache on biopsychosocial status | april 2023-may 2023
  Headache Impact Test (HIT-6™)- A minimum of 36 points and a maximum of 78 points are taken from this scale. The higher the total score obtained from the questionnaire, the worse the quality of life of the participants with headaches.
effect of headache on biopsychosocial status | april 2023-may 2023
  In this form, participants with headaches are asked about the severity of the pain, the frequency, location and duration of the pain, whether there is a family history of headaches, etc.

CONTACTS AND LOCATIONS:
Overall Officials: nezire köse, prof, Study Director — HacettepeUniversity Faculty of Physical Therapy and Rehabilitation
Locations (1):
- Hacettepe Univercity, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stovner Lj, Hagen K, Jensen R, Katsarava Z, Lipton R, Scher A, Steiner T, Zwart JA. The global burden of headache: a documentation of headache prevalence and disability worldwide. Cephalalgia. 2007 Mar;27(3):193-210. doi: 10.1111/j.1468-2982.2007.01288.x. PMID 17381554
- [Background] Bellini B, Arruda M, Cescut A, Saulle C, Persico A, Carotenuto M, Gatta M, Nacinovich R, Piazza FP, Termine C, Tozzi E, Lucchese F, Guidetti V. Headache and comorbidity in children and adolescents. J Headache Pain. 2013 Sep 24;14(1):79. doi: 10.1186/1129-2377-14-79. PMID 24063537
- [Background] Baxter P. ICF: health vs disease. Dev Med Child Neurol. 2004 May;46(5):291. doi: 10.1017/s0012162204000477. No abstract available. PMID 15132257
- See also: The global burden of headache: a documentation of headache prevalence and disability worldwide — https://pubmed.ncbi.nlm.nih.gov/17381554/
- See also: Headache and comorbidity in children and adolescents — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3849985/
- See also: ICF: health vs disease — https://pubmed.ncbi.nlm.nih.gov/15132257/